CLINICAL TRIAL: NCT05773794
Title: Scavenging of Reactive Carbonyl Species by Dietary Flavonoids From Soymilk, Green Tea, and Blueberry in Humans
Brief Title: Scavenging of Reactive Carbonyl Species by Dietary Flavonoids in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina Agriculture & Technical State University (Other)
Responsible Party: Principal Investigator, Shengmin Sang, Distinguished Professor, North Carolina Agriculture & Technical State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 22-0093
Record Dates: First submitted 2023-02-23; First posted 2023-03-17 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Human Health; Reactive Carbonyl Species; Polyphenols
Keywords: dietary flavonoids; Pharmacokinetics; Reactive Carbonyl Species; Polyphenols
MeSH Terms: interventions — Tea; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary flavonoids (soymilk) consumption (Experimental): Week 1: Sixteen healthy volunteers were recruited and instructed to avoid consuming soymilk, green tea, and blueberry products starting one week before the intervention and continuing throughout the entire 3-week study period.
  Week 2: Participants consumed a breakfast including 460 mL of soymilk (or milk) in a single dose. Urine and blood samples were collected at multiple time points over 24 hours, and fecal samples were collected at different time points over 48 hours.
  Week 3: Participants consumed a breakfast including 460 mL of milk (or soymilk) in a single dose. Urine and blood samples were collected at multiple time points over 24 hours, and fecal samples were collected at different time points over 48 hours.
  Interventions: Dietary Supplement: Soymilk, green tea, or blueberry; Dietary Supplement: Control group
- Dietary flavonoids (blueberry) consumption (Experimental): Week 1: Sixteen healthy volunteers were recruited and instructed to avoid consuming soymilk, green tea, and blueberry products starting one week before the intervention and continuing throughout the entire 3-week study period.
  Week 2: Participants consumed a breakfast including 460 mL of blueberry water (or placebo sweet water) in a single dose. Urine and blood samples were collected at multiple time points over 24 hours, and fecal samples were collected at different time points over 48 hours.
  Week 3: Participants consumed a breakfast including 460 mL of placebo sweet water (or blueberry water) in a single dose. Urine and blood samples were collected at multiple time points over 24 hours, and fecal samples were collected at different time points over 48 hours.
  Interventions: Dietary Supplement: Soymilk, green tea, or blueberry; Dietary Supplement: Control group
- Dietary flavonoids (green tea) consumption (Experimental): Week 1: Sixteen healthy volunteers were recruited and instructed to avoid consuming soymilk, green tea, and blueberry products starting one week before the intervention and continuing throughout the entire 3-week study period.
  Week 2: Participants consumed a breakfast including 460 mL of green tea (or water) in a single dose. Urine and blood samples were collected at multiple time points over 24 hours, and fecal samples were collected at different time points over 48 hours.
  Week 3: Participants consumed a breakfast including 460 mL of water (or green tea) in a single dose. Urine and blood samples were collected at multiple time points over 24 hours, and fecal samples were collected at different time points over 48 hours.
  Interventions: Dietary Supplement: Soymilk, green tea, or blueberry; Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Soymilk, green tea, or blueberry — One dose of soymilk, green tea, or blueberry blends (460mL) with breakfast.
Dietary Supplement: Control group — Breakfast with milk or water, without soymilk, green tea, or blueberry blends.

SUMMARY:
This is an interventional study to investigate the formation and pharmacokinetics of reactive carbonyl species adducts of dietary polyphenols (soymilk, green tea, and blueberry) in humans after a single dose of dietary flavonoids.

DETAILED DESCRIPTION:
A crossover design was used. Sixteen healthy volunteers (16 for each study, in total 48) were recruited and asked to avoid the consumption of any soymilk, green tea, and blueberry products starting 1 week before intervention and continuing throughout the entire study for a total of 3 weeks.

On week 2, each of the eight participants received 460 ml of soymilk, green tea, and blueberry in a single dose, and afterward, urine and blood samples at different time points over 24 h and fecal samples at different time points over 48 h were collected. Meanwhile, the other eight participants received breakfast (without any soymilk, green tea, and blueberry) at different time points over 48 h were collected.

On the contrary, on week 3, eight participants who received regular milk or water on week 2 received breakfast only, and eight participants who were used as a control on week 2 received soymilk, green tea, and blueberry. And urine and blood samples at different time points over 24 h, and fecal samples at different time points over 48 h for both groups were collected.

Samples will be analyzed by LC-MS/MS. The Pharmacokinetics of conjugates will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-70 years
2. BMI between 18 and 30
3. Have no known allergy to soy milk
4. Be not taking antibiotics for six months
5. Be not currently taking medication

   1. No taking any prescription drugs
   2. If supplements were taken, flavonoid-enriched supplements (see list below) should be avoided.

      Major brands Notes: All flavonoid-enriched supplements should be avoided. Soy Isoflavones/ tea/blueberry Lipo-Flavonoid Citrus Bioflavonoids Complex Super Flavonoids Super Antioxidants Quercetin Supplement Essential-C and flavonoids Milk Thistle Other flavonoids supplements, including but not limited: Luteolin, Rutin, etc
   3. No any drugs or supplements within three weeks of the experiment
6. Be nonsmoking
7. Have no alcoholic intoxication

   1. No alcoholic addiction
   2. < 3-4 drinks per week (less than 2 glasses (300 mL) per drink)
   3. No alcohol within 3 three weeks of the experiment
8. Have no extended exposure to industrial wastes

Exclusion Criteria:

1. Disease: gout, heart disease, peripheral vascular disease, degenerative kidney, degenerative liver, diabetes, GI disorders, or endocrine disorders
2. Cancer patients

   1. Currently diagnosed cancer patients will be excluded;
   2. Medication free for >2 years could be considered;

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shengmin Sang, PhD, Principal Investigator — NC A&T State University
Locations (1):
- North Carolina Agriculture and Technical State University, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants were asked to avoid the consumption of any soymilk, green tea, and blueberry products one week before the study and continuing throughout the entire study except of the intervention days.
Groups:
- Soymilk Consumption First, Then Placebo: Eight participants consumed 460 mL of soymilk in a single dose on the first intervention and 460 ml of 2% reduced fat milk in a single dose on the second intervention
- Placebo First, Then Soymilk Consumption: Eight participants consumed 460 ml of 2% reduced fat milk in a single dose on the first intervention and 460 ml of soymilk in a single dose on the second intervention
- Green Tea Consumption First, Then Placebo: Seven participants consumed 460 mL of green tea made from 2 servings (4 g) in a single dose on the first intervention and 460 ml water in a single dose on the second intervention
- Placebo First, Then Green Tea Consumption: Nine participants consumed 460 ml water in a single dose on the first intervention and 460 mL of green tea made from 2 servings (4 g) in a single dose on the second intervention
- Blueberry Consumption First, Then Placebo: Eight participants consumed 460 mL of blueberry powder (50 g) in water in a single dose on the first intervention and 460 ml blueberry powder placebo (50 g) in water in a single dose on the second intervention
- Placebo First, Then Blueberry Consumption: Eight participants consumed 460 mL of blueberry powder placebo (50 g) in water in a single dose on the first intervention and 460 mL of blueberry powder (50 g) in water in a single dose on the second intervention
Period: Wash-in Period (1 Week)
Arm/Group | Soymilk Consumption First, Then Placebo | Placebo First, Then Soymilk Consumption | Green Tea Consumption First, Then Placebo | Placebo First, Then Green Tea Consumption | Blueberry Consumption First, Then Placebo | Placebo First, Then Blueberry Consumption
Started | 8 | 8 | 7 | 9 | 8 | 8
Completed | 8 | 8 | 7 | 9 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: First Intervention (1 Day)
Arm/Group | Soymilk Consumption First, Then Placebo | Placebo First, Then Soymilk Consumption | Green Tea Consumption First, Then Placebo | Placebo First, Then Green Tea Consumption | Blueberry Consumption First, Then Placebo | Placebo First, Then Blueberry Consumption
Started | 8 | 8 | 7 | 9 | 8 | 8
Completed | 8 | 8 | 7 | 9 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Wash-out Period (1 Week)
Arm/Group | Soymilk Consumption First, Then Placebo | Placebo First, Then Soymilk Consumption | Green Tea Consumption First, Then Placebo | Placebo First, Then Green Tea Consumption | Blueberry Consumption First, Then Placebo | Placebo First, Then Blueberry Consumption
Started | 8 | 8 | 7 | 9 | 8 | 8
Completed | 8 | 8 | 7 | 9 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Soymilk Consumption First, Then Placebo | Placebo First, Then Soymilk Consumption | Green Tea Consumption First, Then Placebo | Placebo First, Then Green Tea Consumption | Blueberry Consumption First, Then Placebo | Placebo First, Then Blueberry Consumption
Started | 8 | 8 | 7 | 9 | 8 | 8
Completed | 8 | 8 | 7 | 9 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Green Tea Consumption First, Then Placebo: Seven participants consumed 460 mL of green tea made from two servings (4 g) in a single dose on the first intervention and 460 mL of water in a single dose on the second intervention
- Placebo First, Then Green Tea Consumption: Nine participants consumed 460 mL of water in a single dose on the first intervention and 460 mL of green tea made from two servings (4 g) in a single dose on the second intervention
- Blueberry Consumption First, Then Placebo: Eight participants consumed 460 mL of blueberry powder (50 g) in water in a single dose on the first intervention and 460 mL of blueberry powder placebo (50 g) in water in a single dose on the second intervention
- Total: Total of all reporting groups
Arm/Group | Soymilk Consumption First, Then Placebo | Placebo First, Then Soymilk Consumption | Green Tea Consumption First, Then Placebo | Placebo First, Then Green Tea Consumption | Blueberry Consumption First, Then Placebo | Placebo First, Then Blueberry Consumption | Total
Number analyzed (Participants) | 8 | 8 | 7 | 9 | 8 | 8 | 48
Age, Continuous [Mean (Full Range); unit: years] | 35 [23 to 65] | 38.625 [21 to 62] | 47.857 [25 to 59] | 40.11 [25 to 65] | 41.375 [25 to 65] | 44.375 [25 to 65] | 41.0625 [21 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 5 | 4 | 4 | 24
  Male | 4 | 4 | 4 | 4 | 4 | 4 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 1 | 1 | 3 | 2 | 2 | 13
  Black or African American | 0 | 0 | 1 | 0 | 0 | 1 | 2
  White | 4 | 7 | 5 | 6 | 6 | 6 | 34
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 24.89 [20.3 to 27.8] | 26.76 [22 to 33] | 25.21 [18.5 to 36.9] | 23.94 [19.6 to 27.5] | 23.89 [20.56 to 34.39] | 25.25 [20.87 to 28.44] | 25 [18.5 to 36.9]

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary Levels of Reactive Carbonyl Species (RCS) of Soymilk, Green Tea, or Blueberry Over 8 Hours After One Single Dose of Soymilk, Green Tea, or Blueberry Consumption.
Description: Major RCS in urine will be outlined using Liquid chromatography-tandem mass spectrometry (LC-MS). The urinary levels of major RCS over 8 h after one single dose of soymilk, green tea, or blueberry consumption will be quantified using LC-MS.
Time Frame: assessed at 0-2 hours, 2-4 hours, 4-6 hours, and 6-8 hours post-dose
Measure: Mean (Standard Deviation); unit: nmol/mSmo
Groups:
- Soymilk Consumption: Participants consumed 460 mL of soymilk in a single dose. The analysis is to assess the levels of major RCS (MGO) and their major conjugates of polyphenols in human urine.
- Placebo for Soymilk Consumption: Participants consumed 460 ml of 2% reduced fat milk in a single dose. The analysis is to assess the levels of MGO (one of the reactive carbonyl species, RCS) and its major conjugates of polyphenols in human urine.
- Green Tea Consumption: Participants consumed 460 ml of green tea from two serving bags in a single dose. The analysis is to assess the levels of MGO (one of the reactive carbonyl species, RCS) and its major conjugates of polyphenols in human urine.
- Placebo for Green Tea Consumption: Participants consumed 460 ml water in a single dose. The analysis is to assess the levels of MGO (one of the reactive carbonyl species, RCS) and its major conjugates of polyphenols in human urine.
- Blueberry Consumption: Participants consumed 50 g of blueberry powder in 460 ml water in a single dose. The analysis is to assess the levels of MGO (one of the reactive carbonyl species, RCS) and its major conjugates of polyphenols in human urine.
- Placebo for Blueberry Consumption: Participants consumed 50 g of blueberry powder placebo in 460 ml water in a single dose. The analysis is to assess the levels of MGO (one of the reactive carbonyl species, RCS) and its major conjugates of polyphenols in human urine.
Arm/Group | Soymilk Consumption | Placebo for Soymilk Consumption | Green Tea Consumption | Placebo for Green Tea Consumption | Blueberry Consumption | Placebo for Blueberry Consumption
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
nmol/mSmo
  MGO at 0-2 h | 3.71 (0.76) | 4.70 (3.54) | 5.01 (1.40) | 4.98 (0.77) | 7.38 (2.93) | 8.10 (2.72)
  MGO at 2-4 h | 4.41 (0.80) | 3.87 (1.57) | 4.49 (1.06) | 4.79 (0.63) | 7.66 (2.64) | 8.11 (2.24)
  MGO at 4-6 h | 3.37 (0.79) | 2.98 (0.71) | 4.41 (0.66) | 4.60 (0.67) | 5.82 (1.94) | 6.52 (2.13)
  MGO at 6-8 h | 3.23 (1.03) | 3.15 (0.69) | 4.56 (1.14) | 5.06 (1.11) | 4.77 (1.86) | 4.53 (1.17)
Statistical Analysis 1: Comparison: Soymilk Consumption vs Placebo for Soymilk Consumption; Test type: Superiority; p = 0.968, t-test, 2 sided
Statistical Analysis 2: Comparison: Green Tea Consumption vs Placebo for Green Tea Consumption; Test type: Superiority; p = 0.366, t-test, 2 sided
Statistical Analysis 3: Comparison: Blueberry Consumption vs Placebo for Blueberry Consumption; Test type: Superiority; p > 0.05, t-test, 2 sided

2. Primary Outcome: Change in Plasma Levels of Reactive Carbonyl Species (RCS) of Soymilk, Green Tea, or Blueberry Over 4 Hours After One Single Dose of Soymilk, Green Tea, or Blueberry Consumption.
Description: Major RCS in plasma will be outlined using liquid chromatography-tandem mass spectrometry (LC-MS). The major RCS levels in plasma over 4 h after one single dose of soymilk, green tea, or blueberry consumption will be quantified using LC-MS.
Time Frame: assessed at 0 hour, 0.5 hour, 1 hour, 1.5 hours, 2 hours, 3 hours, and 4 hours post-dose
Measure: Mean (Standard Deviation); unit: nM
Groups:
- Soymilk Consumption: Participants consumed 460 mL of soymilk in a single dose. The analysis is to assess the levels of MGO (one of the reactive carbonyl species, RCS) in human plasma.
- Placebo for Soymilk Consumption: Participants consumed 460 ml of 2% reduced fat milk in a single dose. The analysis is to assess the levels of MGO (one of the reactive carbonyl species, RCS) in human plasma.
- Green Tea Consumption: Participants consumed 460 ml of green tea from two serving bags (4 g). The analysis is to assess the levels of MGO (one of the reactive carbonyl species, RCS) in human plasma.
- Placebo for Green Tea Consumption: Participants consumed 460 ml of water. The analysis is to assess the levels of MGO (one of the reactive carbonyl species, RCS) in human plasma.
- Blueberry Consumption: Participants consumed 50 g of blueberry powder in 460 ml water in a single dose. The analysis is to assess the levels of MGO (one of the reactive carbonyl species, RCS) in human plasma.
- Placebo for Blueberry Consumption: Participants consumed 50 g of blueberry powder placebo in 460 ml water in a single dose. The analysis is to assess the levels of MGO (one of the reactive carbonyl species, RCS) in human plasma.
Arm/Group | Soymilk Consumption | Placebo for Soymilk Consumption | Green Tea Consumption | Placebo for Green Tea Consumption | Blueberry Consumption | Placebo for Blueberry Consumption
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
nM
  MGO at 0 h | 388.81 (194.58) | 414.10 (211.59) | 265.62 (90.11) | 266.84 (58.88) | 800.22 (145.41) | 783.50 (151.67)
  MGO at 0.5 h | 349.00 (202.39) | 579.12 (264.45) | 235.66 (99.01) | 245.23 (125.26) | 680.86 (241.39) | 542.16 (184.62)
  MGO at 1.0 h | 508.52 (113.90) | 652.50 (182.36) | 397.41 (227.10) | 434.22 (197.90) | 448.25 (200.51) | 488.45 (323.42)
  MGO at 1.5 h | 281.63 (99.55) | 676.58 (255.80) | 288.82 (124.72) | 276.45 (87.94) | 179.23 (60.95) | 253.73 (190.67)
  MGO at 2.0 h | 403.56 (142.80) | 531.82 (176.33) | 401.58 (193.72) | 414.64 (194.55) | 499.80 (156.25) | 478.71 (152.22)
  MGO at 3.0 h | 253.72 (317.69) | 321.49 (146.08) | 326.86 (165.36) | 403.98 (203.01) | 307.07 (56.13) | 307.85 (92.04)
  MGO at 4.0 h | 252.68 (117.25) | 347.67 (139.16) | 322.85 (130.64) | 342.93 (214.31) | 522.59 (126.55) | 482.44 (191.36)
Statistical Analysis 1: Comparison: Soymilk Consumption vs Placebo for Soymilk Consumption; Test type: Superiority; p = 0.016, t-test, 2 sided
Statistical Analysis 2: Comparison: Green Tea Consumption vs Placebo for Green Tea Consumption; Test type: Superiority; p = 0.11, t-test, 2 sided
Statistical Analysis 3: Comparison: Blueberry Consumption vs Placebo for Blueberry Consumption; Test type: Superiority; p = 0.59, t-test, 2 sided

3. Primary Outcome: Change in Urinary Levels of Reactive Carbonyl Species (RCS) Adducts of Soymilk, Green Tea, or Blueberry Polyphenols Over 24 Hours After One Single Dose of Soymilk, Green Tea, or Consumption.
Description: Major RCS conjugates of polyphenols in urine after soymilk, green tea, or blueberry consumption will be profiled using liquid chromatography-tandem mass spectrometry (LC-MS). The levels of major RCS conjugates in urine over 24 h after soymilk, green tea, or blueberry consumption will be quantified using LC-MS.
Time Frame: 0-2 hours, 2-4 hours, 4-6 hours,6-8 hours, 8-12 hours, and 12-24 hours post-dose
Measure: Mean (Standard Deviation); unit: nmol/mSmo
Groups:
- Soymilk Consumption: Participants consumed 460 mL of soymilk in a single dose. The analysis is to assess the levels of major RCS conjugates of polyphenols in human urine.
- Placebo for Soymilk Consumption: Participants consumed 460 ml of 2% reduced fat milk in a single dose. The analysis is to assess the levels of major RCS conjugates of polyphenols in human urine.
- Green Tea Consumption: Participants consumed 460 ml of green tea from two serving bags in a single dose. The analysis is to assess the levels of major RCS conjugates of polyphenols in human urine.
- Placebo for Green Tea Consumption: Participants consumed 460 ml of water in a single dose. The analysis is to assess the levels of major RCS conjugates of polyphenols in human urine.
- Blueberry Consumption: Participants consumed 50 g of blueberry powder in 460 ml water in a single dose. The analysis is to assess the levels of major RCS conjugates of polyphenols in human urine.
- Placebo for Blueberry Consumption: Participants consumed 50 g of blueberry powder placebo in 460 ml water in a single dose. The analysis is to assess the levels of major RCS conjugates of polyphenols in human urine.
Arm/Group | Soymilk Consumption | Placebo for Soymilk Consumption | Green Tea Consumption | Placebo for Green Tea Consumption | Blueberry Consumption | Placebo for Blueberry Consumption
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
nmol/mSmo
  MGO-EC at 0-2 h | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | 0.042 (0.019) | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified.
  MGO-EC at 2-4 h | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | 0.048 (0.021) | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified.
  MGO-EC at 4-6 h | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | 0.033 (0.013) | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified.
  MGO-EC at 6-8 h | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | 0.018 (0.008) | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified.
  MGO-EC at 8-12 h | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | 0.011 (0.008) | 0.0012 (0.003) | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified.
  MGO-EC at 12-24 h | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | 0.0027 (0.005) | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified. | NA (NA) — The data is below the lower limit of detection and unable to be quantified.
Statistical Analysis 1: Comparison: Green Tea Consumption vs Placebo for Green Tea Consumption; Test type: Superiority; p = 0.0196, t-test, 2 sided
Statistical Analysis 2: Comparison: Soymilk Consumption vs Placebo for Soymilk Consumption; Test type: Superiority; p > 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: Blueberry Consumption vs Placebo for Blueberry Consumption; Test type: Superiority; p > 0.05, t-test, 2 sided

4. Secondary Outcome: Change in Plasma Levels of Reactive Carbonyl Species (RCS) Adducts of Soymilk, Green Tea, or Blueberry Polyphenols Over 24 Hours After One Single Dose of Soymilk, Green Tea, or Consumption.
Description: Liquid chromatography-tandem mass spectrometry will be utilized to assess RCS adducts of soymilk, green tea, or blueberry polyphenols in plasma over 24 hours after one single dose of soymilk, green tea, or blueberry consumption.
Time Frame: 0 hour, 0.5 hour, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, and 24 hours pose dose
Reporting Status: Not Posted, anticipated posting 2026-04

5. Secondary Outcome: Change in Levels of Reactive Carbonyl Species (RCS) Adducts of Soymilk, Green Tea, or Blueberry Polyphenols in Feces Over 48 Hours After One Single Dose of Soymilk, Green Tea, or Consumption.
Description: Major RCS adducts in fecal samples after soymilk, green tea, or blueberry consumption will be profiled. Liquid chromatography-tandem mass spectrometry will be utilized to assess RCS adducts of soymilk, green tea, or blueberry polyphenols in fecal samples.
Time Frame: 0 hour, 24 hours, and 48 hours post-dose
Reporting Status: Not Posted, anticipated posting 2026-04

ADVERSE EVENTS:
Time Frame: 17 days for each intervention.
Groups:
- Soymilk Consumption: Participants consumed 460 mL of soymilk in a single dose.
- Placebo for Soymilk Consumption: Participants consumed 460 mL of 2% reduced fat milk in a single dose.
- Green Tea Consumption: Participants consumed 460 ml of green tea made from 2 servings (4 g) in a single dose.
- Placebo for Green Tea Consumption: Participants consumed 460 ml of water in a single dose.
- Blueberry Consumption: Participants consumed 460 ml of blueberry powder (50 g) in water in a single dose.
- Placebo for Blueberry Consumption: Participants consumed 460 ml of blueberry powder placebo (50 g) in water in a single dose.
Arm/Group | Soymilk Consumption | Placebo for Soymilk Consumption | Green Tea Consumption | Placebo for Green Tea Consumption | Blueberry Consumption | Placebo for Blueberry Consumption
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
N/A. We successfully enrolled 16 participants for each of the three proposed PK studies, with no dropouts during the trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT05773794/Prot_SAP_ICF_000.pdf